CLINICAL TRIAL: NCT01886924
Title: Computer-based MI to Engage Smokers Living With HIV in Tobacco Quitline Treatment
Brief Title: Computer MI for Tobacco Quitline Engagement in Smokers Living With HIV
Acronym: MI-HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA034558
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Smoking Cessation
Keywords: Tobacco; Nicotine; Dependence; Quitline
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Computer MI for Smoking Cessation (Experimental): Brief computer MI intervention to motivate tobacco quitline use
  Interventions: Behavioral: Brief Computer MI for Smoking Cessation
- Nutrition Control (Active Comparator): Computer delivered nutrition education
  Interventions: Behavioral: Nutrition Control

INTERVENTIONS:
Behavioral: Brief Computer MI for Smoking Cessation — Brief computer MI intervention to motivate tobacco quitline use
  Arms: Brief Computer MI for Smoking Cessation
Behavioral: Nutrition Control — Computer delivered nutrition education control condition
  Arms: Nutrition Control

SUMMARY:
The long-term goal of this program of research is to disseminate an effective, brief computer-based intervention that can be readily integrated into HIV treatment settings to motivate tobacco quitline use among smokers living with HIV. The overall objective of this application is to develop this computer intervention, modify it based on initial piloting and feedback, and obtain preliminary data supporting the efficacy of the intervention. This will be accomplished by pursuing three specific aims: 1) to develop and conduct preliminary pilot testing (n=16) of a brief, computer-based intervention intended to motivate tobacco quitline use among cigarette smokers living with HIV (Computer Intervention to Motivate Engagement in Tobacco Quitline treatment; CI-METQ) and to develop and pilot (n=4) a computer-based, time matched nutrition education for PLWH control intervention (NC) equated for the offer of a tobacco quitline referral and 8 weeks of free nicotine patch for those who engage in quitline treatment, 2) to conduct a preliminary smoking cessation, randomized controlled trial (RCT) with 100 people living with HIV (PLWH) who smoke cigarettes, comparing CI-METQ vs. NC, with predictions that CI-METQ relative to NC will result in increased readiness, higher rates of tobacco treatment engagement, more quit smoking attempts and higher rates of 7-day point prevalence abstinence rates at 1-, 3- and 6-month follow-ups. Health-related quality of life over this period will also be examined, and 3) to examine CI-METQ's effects on key mechanisms during the computer session and their associations with tobacco treatment engagement and smoking outcomes at 1- and 3-month follow-ups.

DETAILED DESCRIPTION:
Cigarette smoking is now a leading cause of morbidity and mortality among people living with HIV (PLWH) engaged in highly active antiretroviral therapy (HAART) [2-5]. Between 40-70% of PLWH in the U.S. currently smoke [6-14], in comparison to 20.6% of the general population [15], and tobacco accounted for nearly 25% of all deaths in a multinational cohort of PLWH who used HAART [2]. PLWH who smoke are uniquely vulnerable, moreso than smokers without HIV, to developing cardiovascular [2, 16] and lung [2, 17] diseases, and also are at greater risk than non-smoking PLWH for a multitude of HIV-associated illnesses [3, 5, 18, 19]. Against this backdrop, HIV treatment providers acknowledge the importance of assisting PLWH with smoking cessation, but a significant proportion of them lack confidence, training, and/or time [10, 12, 20]. Very little research on smoking cessation interventions for PLWH has been published, and none has evaluated approaches that could be easily disseminated and integrated into standard HIV care. In this context, a sophisticated, efficacious [ORs, 1.4-1.6 in meta-analyses [21, 22]] tobacco quitline network is now available in every U.S. state via a national quitline portal, 1-800-QUIT-NOW and represents an untapped resource for PLWH. Notably, the most positive findings, to date, for smoking cessation in PLWH have involved telephone counseling delivered by clinical research staff [1], but no existing studies have reported on the efficacy of engaging PLWH with tobacco quitlines or on brief motivational approaches to facilitate this process.

The long-term goal of this research program is to disseminate an effective, brief computer-based intervention that can be readily integrated into community-based, HIV treatment settings to motivate tobacco quitline use among smokers living with HIV. The overall objective of this application, which is the first step in the attainment of our long-term goal, is to develop this computer-based intervention, modify it based on initial piloting and feedback to insure its feasibility and acceptability, and obtain preliminary data supporting the efficacy of the intervention. The rationale for the proposed research is that many smokers living with HIV are interested in quitting smoking, and that by exploring their smoking-related concerns, providing feedback and enhancing self-efficacy, they can become motivated to engage in smoking cessation counseling, utilizing a no-cost, readily available treatment option-their local tobacco quitline. We plan to accomplish the objective of this application by pursuing the following three specific aims:

1. To develop a brief, computer-based intervention, the CI-METQ - Computer Intervention to Motivate Engagement in Tobacco Quitline treatment in PLWH who smoke. Also, to develop a computer-based, time matched nutrition education for PLWH control intervention (NC).

1a. Following the development of the prototype, we will conduct a preliminary pilot test of the CI-METQ with 8 smokers living with HIV, followed by in-depth interviews with each individual to develop an understanding of the strengths and limitations of the intervention. We will then utilize the interview feedback to guide the modification and refinement of the CI-METQ, after which we will repeat the process with another 8 smokers living with HIV.

1b. The data collected from these 16 interviews regarding feasibility, acceptability and barriers that would limit effectiveness will guide the investigators in making the appropriate modifications to finalize the CI-METQ prior to preliminary testing in a small, randomized controlled trial (RCT).

1c. A similar iterative process will occur with 4 PLWH who smoke in developing the NC condition.

2. To conduct a preliminary RCT with 100 smokers living with HIV, comparing CI-METQ to a computer-based, time matched nutrition control (NC) equated for the offer of a tobacco quitline referral and if engaged with quitline, 8 weeks of nicotine patch at no cost. We expect: 2a. CI-METQ relative to NC will result in increased readiness for smoking cessation post-intervention and higher rates of engagement in smoking cessation treatment.

2b. CI-METQ relative to NC will result in a greater proportion of participants making at least one 24 hour quit attempt over the six months post-intervention and in higher rates of 7-day point prevalence abstinence at 1-, 3- and 6- month follow-ups.

2c. To examine the effect of CI-METQ vs. NC on health-related quality of life over 6-month follow-up.

3. To explore potential mechanisms that may underlie the efficacy of CI-METQ: 3a. We will examine CI-METQ's effects on key mechanisms self-reported during the computer session: concerns about cigarette smoking, likelihood of reducing or quitting smoking, health benefits of quitting, and satisfaction with the brief intervention content.

3b. We will examine the associations of these dynamic changes with smoking cessation treatment engagement and smoking outcomes at 1-, 3- and 6-month follow-ups.

With regard to expected outcomes, the work proposed in aims 1 - 3 is expected to result in the development of a brief, computer-based intervention that will produce preliminary data showing increased tobacco quitline utilization and smoking cessation in smokers living with HIV. Such results are expected to have an important positive impact, moving us closer to the long-term goal of dissemination and integration of a cost-effective, CI-METQ into community-based, HIV treatment settings, to motivate tobacco quitline use in PLWH who smoke.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years of age
* current smoker (i.e., at least 10 cigarettes/day)
* HIV seropositive
* English speaking
* reliable access to a telephone (own cellular phone or a landline in their home)
* agreed to be available over the next 6 months.

Exclusion Criteria:

* cognitive impairment sufficient to impair provision of informed consent or study participation
* current use of nicotine replacement therapy (NRT) or other pharmacotherapy for smoking cessation
* use of other tobacco products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Engaged in tobacco cessation treatment since end of treatment intervention | 6 months

SECONDARY OUTCOMES:
Number of quit attempts since last assessment | 6 months

OTHER OUTCOMES:
Point prevalence smoking abstinence - last 7 days from time of assessment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Brown, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States